CLINICAL TRIAL: NCT02468999
Title: Influence of Central Nervous Insulin Action on Insulin Sensitivity of Peripheral Organs in Lean Versus Overweight Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 402/2014B01
Record Dates: First submitted 2015-03-24; First posted 2015-06-11 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Insulin Resistance
Keywords: Intranasal insulin
MeSH Terms: conditions — Insulin Resistance | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- insulin nasal spray (Active Comparator): 160 Units of human insulin as nasal spray
  Interventions: Drug: human insulin
- placebo nasal spray (Placebo Comparator): Nasal spray containing placebo solution
  Interventions: Drug: human insulin

INTERVENTIONS:
Drug: human insulin

SUMMARY:
Research in animals and first experiments in humans indicate that insulin action in the brain regulates peripheral insulin sensitivity. One major organ might be the liver. Previous studies in humans showed that the human brain is an insulin sensitive organ in lean but not in overweight/obese persons. Therefore, this study will include lean versus overweight/obese persons.

In this study, insulin action will be introduced by intranasal insulin administration in lean and overweight humans. As a control, placebo spray will be administered. To mimick the known spill over of small amounts of intranasal insulin into circulation, a small bolus of insulin will be administered over 15 minutes following placebo spray application.

Peripheral insulin sensitivity will be assessed by hyperinsulinemic-euglycemic glucose clamp and glucose uptake and endogenous glucose production will be assessed by tracer dilution technique. Autonomous nervous system activity will be addressed by heart rate variability. Involved brain areas will be addressed by fMRI before and after nasal insulin application.

ELIGIBILITY:
Inclusion Criteria:

* Male volunteers (lean or overweight/obese)
* HbA1c <6.0%
* Age between 18 and 40 years
* healthy as assessed by physician
* Understanding the explanations about the study and instructions

Exclusion Criteria:

* non-removable metal parts in or on the body
* Persons with reduced temperature sensation and / or increased sensitivity to warming of the body
* Cardiovascular disease can not be excluded, such as evident coronary heart disease, congestive heart failure NYHA greater than 2, history of coronary artery disease
* History of stroke
* Persons with a hearing disorder or increased sensitivity to loud noises
* People with claustrophobia
* Subjects in which less than 3 months have passed since surgery
* Simultaneous participation in other studies
* Acute disease or infection within the last 4 weeks
* Neurological and psychiatric disorders
* Subjects with hemoglobin Hb <13g / dl
* Heparin-induced thrombocytopenia people with a (HIT) in prehistory
* Allergies to any of the used solutions/devices

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in glucose infusion rate during hyperinsulinemic euglycemic glucose clamp from before to after nasal spray application in lean persons | Change from 70-90 min (before spray) to 170-210 min and to 280-300 min
Change in endogenous glucose production from before to after nasal spray application in lean persons | Change from 70-90 min (before spray) to 170-210 min and to 280-300 min
  Will be assessed by tracer dilution technique.
Differences in insulin response between lean and overweight persons | up to 210 minutes post nasal spray administration
  Will be assessed as plasma insulin and C-peptide concentrations.

SECONDARY OUTCOMES:
Autonomous nervous system activity | baseline, 70-90 min, 170-210 min and 280-300 min
  Will be assessed by analysis of heart rate variability.
Regional brain insulin sensitivity | 30 min
  Will be assessed on an additional study day by fMRI before and after intranasal insulin administration

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Fritsche, Prof. Dr., Principal Investigator — University Hospital Tuebingen
Locations (1):
- University of Tuebingen, Department of Internal Medicine IV, Tübingen, Germany

REFERENCES:
- [Derived] Heni M, Wagner R, Kullmann S, Gancheva S, Roden M, Peter A, Stefan N, Preissl H, Haring HU, Fritsche A. Hypothalamic and Striatal Insulin Action Suppresses Endogenous Glucose Production and May Stimulate Glucose Uptake During Hyperinsulinemia in Lean but Not in Overweight Men. Diabetes. 2017 Jul;66(7):1797-1806. doi: 10.2337/db16-1380. Epub 2017 Feb 7. PMID 28174292